CLINICAL TRIAL: NCT02426593
Title: Collection of Anatomical and Reference Data for Development of a Novel Non-Invasive Lung Hydration Status Technology
Status: Completed | Type: Observational
Sponsor: Intersection Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-000060
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: CHF; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects without heart failure
  Interventions: Device: IMED-4

INTERVENTIONS:
Device: IMED-4 — Non-invasive novel lung hydration status sensor.

SUMMARY:
This study will be conducted to collect anatomical data in an ambulatory healthy population to aid in the development of a novel non-invasive technology to assess changes in lung hydration status. It will also help in developing reference ranges of lung hydration status in healthy subjects and their associated changes with time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 30 years of age
* Subjects who are ambulatory not requiring assistance for ambulation
* Subjects who have been informed of the nature of the study and agree to its provisions and have provided written informed consent as approved by the IRB

Exclusion Criteria:

* Subjects with an active implantable medical device not cleared for use with the IMED-4 in the IMED- 4 Investigators Brochure.
* Subjects who are pregnant or lactating or who have been pregnant within the past three months
* Subjects who have a measured temperature of >38° C at the time of screening
* Subjects who have tattoos and/or non-intact skin on the back in the electrode patch placement region
* Subjects who have had a past serious allergic reaction to adhesives
* Patients who decline to have their backs photographed with the IMED-4 device in position
* Subjects who have poor general physical/mental health that, in the opinion of the investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, incarceration, shortened life expectance, etc.)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the general population using various media advertising as well as through a site database. Potential subjects aged older than 30 will be recruited for a telephone interview. If they qualify based on a very brief screening interview regarding their suitability as a participant, and they are interested in participating, they will be scheduled to visit the Intersection Medical, Inc., corporate office. If they decline to participate, no further contact will be initiated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Data Collection | 12 months
  The primary endpoint is successful IMED-4 recordings at multiple timepoints from one hundred (100) unique subjects. A recording will be considered successful if it meets IMED-4 recording quality indicators.

CONTACTS AND LOCATIONS:
Locations (1):
- Intersection Medical Inc., Carlsbad, California, United States